CLINICAL TRIAL: NCT06742645
Title: The Use of Brief Motivational Interviewing in Community Health Centers. Controlled Trial on Quality of Life and Perceived Health Status
Brief Title: The Use of Brief Motivational Interviewing in Community Health Centers.
Acronym: BMICHC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24014 - 81-2024-SPER-AUSLBO
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Healthy Subjects
Keywords: Motivational Interviewing
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: INTERVENTION The health workers of the Borgo Reno Community House perform the outpatient visit and after having identified the health problems they propose a possible treatment. Subsequently, the citizen included in the study is subjected to the intervention, short motivational interview (BMI). By putting the relationship, listening, assertive communication, motivation and direct involvement of the patient in the treatment path in the foreground, the trained workers conduct the BMI to motivate the users of the various services to improve their lifestyles. Objectives to be achieved within six months will be agreed upon. The short motivational interview lasts approximately 15 minutes COMPARISON The health workers of the Navile Community House perform the outpatient visit and after having identified the health problems they propose a possible treatment. The users belonging to the control arm will complete the SF-36 questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Community House Borgo Reno (Experimental): The health workers of the Borgo Reno Community House perform the outpatient visit and after having identified the health problems they propose a possible treatment. Subsequently, the citizen included in the study is subjected to the intervention, short motivational interview (BMI). By putting the relationship, listening, assertive communication, motivation and direct involvement of the patient in the treatment path in the foreground, the trained workers conduct the BMI to motivate the users of the various services to improve their lifestyles. Objectives to be achieved within six months will be agreed upon. The short motivational interview lasts approximately 15 minutes
  Interventions: Behavioral: Brief Motivational Interviewing
- Community House Navile (Active Comparator): The health workers of the Navile Community House perform the outpatient visit and after having identified the health problems they propose a possible treatment. The users belonging to the control arm will complete the SF-36 questionnaire Send feedback
  Interventions: Behavioral: Standard of Care (SOC)

INTERVENTIONS:
Behavioral: Brief Motivational Interviewing — Brief Motivational Interviewing (BMI), the object of the training and of the present research study, is an interview methodology that includes the intervention on the motivation to change of subjects with risky behaviors for their health, in order to obtain changes in their lifestyle and maintain correct behaviors for health over time (1). The BMI is mainly based on the Transtheoretical Model of Change by Di Clemente CC. and Prochaska JO (2).
  In particular, the BMI has been defined by its creators, Miller and Rollnick, as "a collaborative style of conversation aimed at strengthening motivation and commitment to change" (3), both through defined attitudes, strategies and techniques, and through the exploration of ambivalence or internal fracture, which together with availability and a sense of self-efficacy (4) provides a framework of personal motivation.
  Arms: Community House Borgo Reno
Behavioral: Standard of Care (SOC) — Standard of Care (SOC) - The health workers of the Navile Community House carry out the outpatient visit and after having identified the health problems they propose a possible treatment. The users belonging to the control arm will complete the SF-36 questionnaire
  Arms: Community House Navile

SUMMARY:
The research project aims to detect the effect of the Brief Motivational Interview (BMI) on the motivation to change risky behaviors and the adoption of healthy lifestyles by citizens attending Community Health Centers (CdC). The controlled, multicenter, prospective design study involves the enrollment of 304 people, with 152 at the Borgo Reno CdC and 152 at the Navile CdC.

DETAILED DESCRIPTION:
The study will include 152 citizens who use the services of the Borgo Reno Community Health Center and 152 citizens from the Navile Community Health Center. Eligible participants will be identified with the help of specialist medical staff and nursing staff at the facility. Once an eligible participant is identified, the Brief Motivational Interview (BMI) can be conducted during regular institutional activities (if the operator on duty at that time is trained to conduct the BMI and after obtaining informed consent and completing the SF-36 questionnaire) or by scheduling an appointment with the nursing and/or facility staff for a dedicated BMI clinic.

Students from the degree courses in "Psychology," "Human Nutrition, Wellness, and Health," and "Wellness, Sport, and Health," who are appropriately trained and authorized, will contribute to the research study by providing all necessary information. Participants in the experimental group who are given an appointment will sign the informed consent for participation and consent for the processing of personal and sensitive data. They will also receive a letter for their general practitioner explaining the study procedures. Inclusion and exclusion criteria will be assessed. If the criteria are met, the citizen will be included in the study.

Citizens enrolled at the Borgo Reno Community Health Center will be assigned to the experimental group (with intervention), while those enrolled at the Navile Community Health Center will be part of the control group (without intervention). A clinic will be dedicated to this study, where professionals (specialist/home nursing staff, dietitians, physiotherapists, IFeC) from the Community Health Center who have received training from the CCM course on Brief Motivational Interviewing will conduct the sessions.

ELIGIBILITY:
Inclusion Criteria:

* first visit to the Cardiology or Endocrinology/Diabetology or Rheumatology or Basic Dietetics services or other medical specialties of the Borgo-Reno or Navile Community Home or referred to them.
* resident in the AUSL of Bologna
* age ≥18 years

Exclusion Criteria:

* second or more visits to the Cardiology or Endocrinology/Diabetology or Rheumatology or Basic Dietetics services, or other medical specialties of the Borgo-Reno or Navile Community House or referred to them.
* first visit to a service not indicated in the inclusion criteria
* not resident in the territory of the AUSL of Bologna
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | From enrollment to the end of treatment at 6 MONTHS
  The 36-item Short Form Health Survey (SF-36) is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Sanità Pubblica, Bologna, IT, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Ghizzardi G, Arrigoni C, Dellafiore F, Vellone E, Caruso R. Efficacy of motivational interviewing on enhancing self-care behaviors among patients with chronic heart failure: a systematic review and meta-analysis of randomized controlled trials. Heart Fail Rev. 2022 Jul;27(4):1029-1041. doi: 10.1007/s10741-021-10110-z. Epub 2021 Apr 17. PMID 33866487
- [Background] Pedamallu H, Ehrhardt MJ, Maki J, Carcone AI, Hudson MM, Waters EA. Technology-Delivered Adaptations of Motivational Interviewing for the Prevention and Management of Chronic Diseases: Scoping Review. J Med Internet Res. 2022 Aug 9;24(8):e35283. doi: 10.2196/35283. PMID 35943775
- [Background] Rogers CR. A theory of therapy, personality and interpersonal relationships as developed in the client-centered framework. In: Koch S. (ed). Psychology: a study of a science, vol. III. Formulations of the person in the social context. McGraw Hill, New York, 1959.
- [Background] Bandura A., Self-efficacy mechanism in human agency. American Psychologist, 1982; 37: 122-47
- [Background] Miller WR, Rollnick S. Motivational Interviewing. Helping people change. Guilford Press, New York, 1991.
- [Background] Prochaska JO. Di Clemente CC. Transtheorical therapy: toward a more integrative model of change. Psychotherapy, theory, research and practice 1982.
- [Background] Britt E, Hudson SM, Blampied NM. Motivational interviewing in health settings: a review. Patient Educ Couns. 2004 May;53(2):147-55. doi: 10.1016/S0738-3991(03)00141-1. PMID 15140454